CLINICAL TRIAL: NCT05724459
Title: The Effect of Peer Education on Stem Cell Donation in Nursing Students on Their Knowledge and Attitudes About Being a Hematopoietic Stem Cell Donor
Brief Title: The Effect of Peer Education on Stem Cell Donation in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Prof., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Peer Education on Stem Cell
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Nursing Students
Keywords: Nursing Students; Stem Cell Transplantation; Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Education Group (Experimental): Training on stem cell transplantation for a total of 12 hours, two days a week for three weeks, two lesson hours a day (60 min. + 60 min.)
  Interventions: Other: Peer education
- Control Group (No Intervention)

INTERVENTIONS:
Other: Peer education — Training on stem cell transplantation for a total of 12 hours, two days a week for three weeks, two lesson hours a day (60 min. + 60 min.)
  Arms: Peer Education Group

SUMMARY:
The aim of the study is to determine the effect of peer education on stem cell donation in nursing students on their knowledge and attitudes towards being a stem cell donor. This study is a randomized-controlled experimental design study. The dependent variable of the study is the knowledge and attitudes of nursing students towards being a stem cell donor. The independent variable is peer education on stem cell donation. The research will be carried out with nursing students studying at the Nursing Department of a university located in Istanbul. The universe of the research will be all students (N= 320) studying in the Department of Nursing in the 2022-2023 academic year. The sample of the research will consist of our friends from the nursing department who volunteered to participate in the research. In the power analysis to calculate the sample size, the sample size of the study was calculated as at least 88 for each group, with an effect size of 0.50, a margin of error of 5%, and a power of 95%. However, it was aimed to reach 100 students for each group, in case the participants were withdrawn from the study during the research and education process and the sample size could not be reached. Introductory Information Form and Stem Cell Transplant Information Form will be used to collect data. The data in the research will be collected in two stages. In the first stage, peer educators will be trained and evaluated by our consultant, who is a project internal medicine nursing specialist. In the second stage, peer educators will train and evaluate peer students. After our students studying in the nursing department who meet the sampling criteria are informed about the study, informed consent forms will be signed by face-to-face interview. Peer students will be randomly assigned to the intervention (100 people) and control (100 people) groups according to the randomization list prepared in advance. Peer educators will train nursing students in the intervention group with the peer education model. No application will be made to the control group. Pre-test data will be obtained by applying the measurement tools to both groups at the beginning of the study. After the intervention group is trained, the Stem Cell Transplant Information Form will be filled in at the first follow-up at the 3rd month and at the second follow-up at the 6th month. The follow-up of the students in the control group will be done in a similar way. The results will be analyzed with the SPSS program. In the analysis of socio-demographic data, number, percentage, mean, median (median), standard deviation will be used. In the data showing normal distribution, Independent Samples T test will be used for comparisons between two groups, one of the parametric tests, and One Way ANOVA test will be used if there are 3 or more groups. For data that does not show normal distribution, the Mann-Whitney U test will be used for comparisons between two groups, one of the non-parametric tests, and the Kruskall Wallis test if there are 3 or more groups. As a result of this study, the effect of peer education and training on the stem cell donation knowledge levels of nursing students and their attitudes towards stem cell donation will be evaluated.

DETAILED DESCRIPTION:
Hematopoietic stem cells (HSC) are cells that can be produced in adults with special methods and with the help of certain growth factors and can turn into blood cells. The collection of stem cells from the individual or from a different person compatible with the tissue group and giving them to the patient after the preparation regimen is defined as peripheral hematopoietic stem cell transplantation, and the delivery of the product collected by aspiration from the posterior iliac bone with special aspiration needles under general anesthesia to the patient is defined as bone marrow transplantation (Suluhan et al. et al., 2016). Hematopoietic stem cell transplantation (HSCT) is the most commonly used stem cell therapy today. Target cells are obtained from bone marrow, peripheral blood or umbilical cord blood (Zakrzewski et al., 2019). HSCT is very important in the treatment of many diseases that may result in death, some types of cancer (such as leukemia, bone marrow cancer, lymphoma) and congenital blood diseases. In addition, important developments have been made in stem cell therapy for the treatment of many neurological diseases such as stroke due to spinal cord injuries and cerebrovascular occlusion, as well as progressive diseases such as Alzheimer's and Parkinson's (Barriga et al., 2012). Anyone who is healthy between the ages of 18 and 50 can be a donor for stem cell donation. Stem cells collected from the blood in the peripheral body circulation are the most commonly used donation method. Another donation method is bone marrow (Dinç & Şahin, 2010).

It is very important to raise awareness of the society about stem cell donation. Many volunteers, who are stem cell donors, are needed for the treatment of many patients awaiting transplantation. According to World Bone Marrow Donor Association (WMDA) data, there are 37,179,232 donors and 800,090 cord blood units registered in bone marrow and cord blood banks in 55 different member countries (https://statistics.wmda.info). According to the data of the Turkish Stem Cell Coordination Center (TÜRKÖK), 766,000 stem cell samples were registered in 2020. However, more hematopoietic stem cell donation is needed. The lack of information, misinformation, unfounded fears and concerns about stem cell donation in the general population cause the needed number of donors not to be reached (Savran, 2021).

In studies conducted in our country, it is reported that many people in the society have low level of knowledge about stem cells. In their study, Dinç and Şahin (2010) examined the knowledge and approaches of student nurses / midwives about stem cells and cord blood, it was found that nearly half of the participants had an idea about stem cells and cord blood, but their level of knowledge was insufficient. It was determined that 24% of them obtained information from the media and 17% from courses. Although many national and international activities are carried out to increase the donor rate, the donor rates of active and healthy people in the 18-25 age group are not sufficient. In the donor analyzes published by WMDA, donations made by the 18-25 age group constitute 14.3% of all donations (WMDA Global Trend Report, 2018). In a web-based study conducted by Kwok et al. in Hong Kong to determine the factors affecting being a hematopoietic stem cell donor; A significant relationship was found between age, education level, HKHN knowledge score and donation intention (Kwok et al. 2015). Sikora et al.'s study on university students in Lublin revealed that reluctance to donate was due to lack of knowledge and fear of being harmed in the younger group (Sikora et al. 2014). As a result of another study conducted in America; The students stated that there is a lack of knowledge and they are afraid of the side effects that may occur after the transplant. Lack of knowledge in students causes prejudices about donation (Narayanan et al. 2016). As it can be understood from the results of the study, the lack of knowledge of young people about stem cell donation prevents people from being a donor. In order to increase social sensitivity and awareness; It is important to investigate, examine and examine how healthcare professionals and nursing students, who are health worker candidates, evaluate stem cell studies (Suluhan et al., 2016).

The peer education model, which has a wide place among the new education methods, was created based on the fact that young people interact well with their peers and identify with each other, and in this model, people with similar status train and guide each other as knowledge and skills through activities such as seminars, case presentations, practices and discussions. (Unver and Akbayrak, 2013; Şenyuva and Akince, 2020). Social interaction in peer education method; Sharing the cognitive load is very important because those who know better share what they know with those who do not know, and internalize what they have learned within the peer group. Peer trainers are very effective in developing and encouraging healthy behavior (Şenyuva & Akince, 2020). With this training, the health status of both themselves and the society can be protected and improved by ensuring that young people acquire accurate information about many different fields, especially sensitive, private and taboo subjects. From this point of view, it is expected that the peer education given to nursing students about stem cell donation will contribute positively to their knowledge and attitudes towards being a stem cell donor. It is thought that this study will contribute to studies evaluating the effect of education on stem cell donation and knowledge level, which are limited in the literature (Kaya et al., 2015; Karakaçan, 2020). The aim of the study is to determine the effect of peer education on stem cell donation in nursing students on their knowledge and attitudes towards being a stem cell donor. This study is a randomized-controlled experimental design study. The dependent variable of the study is the knowledge and attitudes of nursing students towards being a stem cell donor. The independent variable is peer education on stem cell donation. The research will be carried out with nursing students studying at the Nursing Department of a university located in Istanbul. The universe of the research will be all students (N= 320) studying in the Department of Nursing in the 2022-2023 academic year. The sample of the research will consist of our friends from the nursing department who volunteered to participate in the research. In the power analysis to calculate the sample size, the sample size of the study was calculated as at least 88 for each group, with an effect size of 0.50, a margin of error of 5%, and a power of 95%. However, it was aimed to reach 100 students for each group, in case the participants were withdrawn from the study during the research and education process and the sample size could not be reached. Introductory Information Form and Stem Cell Transplant Information Form will be used to collect data. The data in the research will be collected in two stages. In the first stage, peer educators will be trained and evaluated by our consultant, who is a project internal medicine nursing specialist. In the second stage, peer educators will train and evaluate peer students. After our students studying in the nursing department who meet the sampling criteria are informed about the study, informed consent forms will be signed by face-to-face interview. Peer students will be randomly assigned to the intervention (100 people) and control (100 people) groups according to the randomization list prepared in advance. Peer educators will train nursing students in the intervention group with the peer education model. No application will be made to the control group. Pre-test data will be obtained by applying the measurement tools to both groups at the beginning of the study. After the intervention group is trained, the Stem Cell Transplant Information Form will be filled in at the first follow-up at the 3rd month and at the second follow-up at the 6th month. The follow-up of the students in the control group will be done in a similar way. The results will be analyzed with the SPSS program. In the analysis of socio-demographic data, number, percentage, mean, median (median), standard deviation will be used. In the data showing normal distribution, Independent Samples T test will be used for comparisons between two groups, one of the parametric tests, and One Way ANOVA test will be used if there are 3 or more groups. For data that does not show normal distribution, the Mann-Whitney U test will be used for comparisons between two groups, one of the non-parametric tests, and the Kruskall Wallis test if there are 3 or more groups. As a result of this study, the effect of peer education and training on the stem cell donation knowledge levels of nursing students and their attitudes towards stem cell donation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Willing to participate in the study,
* A permanent student in the nursing department and
* Students who do not have any communication problems will be included in the study.

Exclusion Criteria:

* Any communication barriers
* Students who do not volunteer to participate in the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | 1. day
  It consists of two parts. The first part includes demographic information such as age, education level, income level, occupation, and length of work in the profession. In the second part, there are questions about their views on stem cell donation. It covers questions about students' awareness of stem cells, whether they are a stem cell donor in their environment, whether they give stem cell donation samples, and their opinions and attitudes on this subject.
Stem Cell Transplant Information Form | 1. day
  It was developed by Çiçek and Dinç in 2022 (Çiçek and Dinç, 2022). There are knowledge level questions about stem cell donation. In this section, 1) General information about stem cells, 2) Stem cell collection by peripheral method (blood, apheresis process), 3) Stem cell collection from bone marrow 4) Information questions about stem cell donation. Incorrect answers to questions measuring the level of knowledge; 2, 15, 19, 20, 21, 22, 23, correct questions are indicated in 1, 3-14, 16-18, 24,25. The knowledge score obtained from the test is a minimum of 0 and a maximum of 20 points.
Stem Cell Transplant Information Form | 90th day
  It was developed by Çiçek and Dinç in 2022 (Çiçek and Dinç, 2022). There are knowledge level questions about stem cell donation. In this section, 1) General information about stem cells, 2) Stem cell collection by peripheral method (blood, apheresis process), 3) Stem cell collection from bone marrow 4) Information questions about stem cell donation. Incorrect answers to questions measuring the level of knowledge; 2, 15, 19, 20, 21, 22, 23, correct questions are indicated in 1, 3-14, 16-18, 24,25. The knowledge score obtained from the test is a minimum of 0 and a maximum of 20 points.
Stem Cell Transplant Information Form | 180th day
  It was developed by Çiçek and Dinç in 2022 (Çiçek and Dinç, 2022). There are knowledge level questions about stem cell donation. In this section, 1) General information about stem cells, 2) Stem cell collection by peripheral method (blood, apheresis process), 3) Stem cell collection from bone marrow 4) Information questions about stem cell donation. Incorrect answers to questions measuring the level of knowledge; 2, 15, 19, 20, 21, 22, 23, correct questions are indicated in 1, 3-14, 16-18, 24,25. The knowledge score obtained from the test is a minimum of 0 and a maximum of 20 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No